CLINICAL TRIAL: NCT06253195
Title: A Phase 1a/1b Study Investigating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Antitumor Activity of the CDK4 Inhibitor BGB-43395, Alone or as Part of Combination Therapies in Chinese Patients With Advanced or Metastatic HR+/HER2- Breast Cancer and Other Solid Tumors
Brief Title: BGB-43395 Alone or as Part of Combination Therapies in Chinese Participants With HR+/HER2- Breast Cancer and Other Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BGB-43395-102; CTR20240674 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor; Hormone-receptor-positive Breast Cancer; Breast Cancer; Metastatic Breast Cancer; Hormone Receptor Positive Malignant Neoplasm of Breast; HER2-negative Breast Cancer
Keywords: advanced solid tumor; metastatic solid tumor; BGB-43395; breast cancer; HR+/HER2- breast cancer; hormone receptor positive breast cancer
MeSH Terms: conditions — Neoplasm Metastasis; Breast Neoplasms | interventions — Fulvestrant; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1a: Dose Escalation (Experimental): Sequential cohorts of increasing dose levels of BGB-43395 will be evaluated as monotherapy and in combination with either fulvestrant or letrozole.
  Interventions: Drug: BGB-43395; Drug: Fulvestrant; Drug: Letrozole
- Phase 1b: Dose Expansion (Experimental): The recommended dose for expansion (RDFE) for BGB-43395 in combination with fulvestrant from Phase 1a will be evaluated in HR+ breast cancer and selected tumor cohorts.
  Interventions: Drug: BGB-43395; Drug: Fulvestrant

INTERVENTIONS:
Drug: BGB-43395 — Administered orally.
Drug: Fulvestrant — Administered via intramuscular injection.
Drug: Letrozole — Administered orally.
  Arms: Phase 1a: Dose Escalation

SUMMARY:
This is an open-label, multicenter, phase 1a/1b clinical study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary antitumor activity of BGB-43395, a cyclin-dependent kinase 4 (CDK4) inhibitor, as monotherapy or in combination with fulvestrant, letrozole, or other combination partners in Chinese participants with hormone receptor positive (HR+) and human epidermal growth factor 2 negative (HER2-) breast cancer (BC) and other advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1a (Dose Escalation): Participants with histologically or cytologically confirmed locally advanced or metastatic solid tumors associated with CDK4 dependency, including HR+/HER2- breast cancer. Participants must have received prior standard-of-care therapies for their disease, unless the therapy is not available or not tolerated, or is determined not appropriate based on the investigator's judgment.
* Phase 1b (Dose Expansion): Participants with selected solid tumors including locally advanced or metastatic HR+/HER2- breast cancer.
* Female participants with metastatic HR+/HER2- breast cancer will be required to have ovarian function suppression using gonadotropin-releasing hormone (GnRH) agonists such as goserelin or be postmenopausal.
* Male participants with HR+/HER2- breast cancer will be required to have gonadal suppression using GnRH agonists when being treated with letrozole or fulvestrant.
* Patients must have ≥1 measurable lesion per RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1.
* Adequate organ function without symptomatic visceral disease.

Exclusion Criteria:

* Prior therapy selectively targeting CDK4 (prior CDK4/6 inhibitor therapy is permitted).
* Known leptomeningeal disease or uncontrolled untreated brain metastasis.
* Any malignancy ≤ 3 years before the first dose of study drug(s) except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated with curative intent (eg, resected basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix or breast).
* Uncontrolled diabetes.
* Infection requiring systemic antibacterial, antifungal, or antiviral therapy ≤ 28 days before the first dose of study drug(s), or symptomatic COVID-19 infection. Patients receiving prophylactic antibiotics (eg, for prevention of urinary tract infection, chronic obstructive pulmonary disease, or for dental extraction) are eligible. Patients who have recovered from symptomatic COVID-19 infection can be rescreened for this study.
* Untreated chronic hepatitis B or active hepatitis C infection.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-10-26 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to approximately 30 months
  Number of participants with AEs and SAEs including findings from physical examinations, electrocardiograms (ECGs), and laboratory assessments as needed, and that meet protocol-defined dose-limiting toxicity (DLT) criteria.
Phase 1a: Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD) of BGB-43395 | Up to approximately 30 months
  MTD is defined as the highest dose evaluated for which estimated toxicity rate is the closest to the target toxicity rate. MAD is defined as the highest dose administered if MTD is not reached.
Phase 1a: Recommended Dose for Expansion (RDFE) of BGB-43395 | Up to approximately 30 months
  RDFE of BGB-43395 alone or as part of combination therapies will be determined based upon the MTD or MAD.
Phase 1b: Objective Response Rate (ORR) | Up to approximately 30 months
  ORR is defined as the percentage of participants who have confirmed complete response (CR) or partial response (PR) as assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

SECONDARY OUTCOMES:
Phase 1a: ORR | Up to approximately 30 months
  ORR is defined as the percentage of participants who have confirmed CR or PR assessed by the investigator using RECIST v1.1.
Phase 1b: Progression-Free Survival (PFS) | Up to approximately 30 months
  PFS is defined as the time from the date of the first dose of study drug(s) to the date of the first documentation of progressive disease assessed by the investigator using RECIST v1.1 or death, whichever occurs first.
Phase 1b: Number of Participants with AEs and SAEs | Up to approximately 30 months
  Number of participants with AEs and SAEs including findings from physical examinations, ECGs, and laboratory assessments as needed.
Phase 1a and 1b: Duration of Response (DOR) | Up to approximately 30 months
  DOR is defined as the time from the first determination of an objective response by the investigator using RECIST v1.1 until the first documentation of disease progression or death, whichever occurs first.
Phase 1a and 1b: Time to Response (TTR) | Up to approximately 30 months
  TTR is defined as the time from the date of the first dose of study drugs to the date of the first determination of objective response that is confirmed by a subsequent response as assessed by the investigator using RECIST v1.1.
Phase 1b: Disease Control Rate (DCR) | Up to approximately 30 months
  DCR is defined as the percentage of participants with best overall response of CR, PR, or stable disease assessed by the investigator using RECIST v1.1.
Phase 1b: Clinical Benefit Rate (CBR) | Up to approximately 30 months
  CBR is defined as the percentage of participants with best overall response of confirmed CR, PR, or stable disease lasting ≥ 24 weeks.
Phase 1a: Observed plasma maximum concentration (Cmax) of BGB-43395 and its metabolite | From Cycle 1 Day 1 up to Cycle 7 Day 1 (each cycle is 28 days)
Phase 1a: Observed plasma trough concentration (Ctrough) of BGB-43395 and its metabolite | From Cycle 1 Day 1 up to Cycle 7 Day 1 (each cycle is 28 days)
Phase 1a: Area under the concentration-time curve (AUC) of BGB-43395 and its metabolite | From Cycle 1 Day 1 up to Cycle 7 Day 1 (each cycle is 28 days)
Phase 1a: Half-life (t1/2) of BGB-43395 and its metabolite | From Cycle 1 Day 1 up to Cycle 7 Day 1 (each cycle is 28 days)
Phase 1b: Plasma concentrations of BGB-43395 and its metabolite | From Cycle 1 Day 1 up to Cycle 5 Day 1 (each cycle is 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (7):
- China (7):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat Sen Memorial Hospital, Sun Yat Sen University (South), Guangzhou, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/